CLINICAL TRIAL: NCT00719433
Title: Functional Recovery in Stroke Patients With Task-Specific Robot-Aided Arm Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Sensory Motor Systems Lab, ETH Zurich (Unknown); Balgrist University Hospital (Other); Reha Rheinfelden (Other); Zuercher Hoehenklinik Wald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNF ARMin III -1; SNF 325200-120621; EK-39/2007
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Stroke; Upper Extremity Paresis
Keywords: stroke; chronic; rehabilitation; robot therapy; arm therapy
MeSH Terms: conditions — Stroke; Paresis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: robot therapy (ARMin)
- 2 (Active Comparator)
  Interventions: Other: conventional therapy

INTERVENTIONS:
Device: robot therapy (ARMin) — therapy of the affected arm with a robot for eight weeks, three times weekly for one hour
  Arms: 1
Other: conventional therapy — physical and occupational therapy of the affected arm for eight weeks, three times weekly for one hour
  Arms: 2

SUMMARY:
The goal of this study is to determine whether task-oriented, robot-aided therapy is more effective than conventional physical and occupational therapy at promoting functional recovery of the affected arm in chronic hemiparetic stroke patients.

DETAILED DESCRIPTION:
Robotic therapy will be performed with ARMin, which is a robotic arm exoskeleton that permits 3D movements of both proximal and distal arm joints. Combined with an audiovisual display, this device allows virtual training of Activities of Daily Living (ADL) and therapeutic gaming. A patient-responsive controller enables the assistance of the device only as needed. Chronic stroke patients (>6 months post stroke) will be randomly assigned to either an experimental or a control group. The experimental group will perform task-related intensive therapy with the support of ARMin. Therapists will treat the patients of the control group with standard motor relearning therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or more
* first-ever stroke (hemorrhagic or ischemic), verified by brain imaging
* stroke more than six months prior to the study
* termination of conventional therapy and stable recovery stage (outpatients)
* moderate to severe motor impairment of the arm (upper limb portion of FMA score between 8 and 38)
* ability to sit in a chair without any additional support and without leaning on the back rest
* written informed consent signed by the subject (or an authorized representative)

Exclusion Criteria:

* Excessive spasticity of the affected arm (mAS ≥ 3)
* any serious medical or psychiatric illness
* participation in any clinical investigation within 4 weeks prior to the start of this study
* anticipated need for any major surgery during the study
* women known to be pregnant or lactating
* Orthopedic, rheumatologic or other disease restricting movements of the paralyzed upper extremity
* shoulder subluxation (palpatory > 2 fingers)
* diseased or damaged skin at the paralyzed arm
* inability to communicate effectively with the neurological examiner such that the validity of the patient's data could be compromised
* cyber sickness
* pace-maker or other implanted electric devices
* body weight > 120kg
* serious cognitive deficits and aphasia preventing the performance of the ARMin treatment
* participation in any therapeutic treatment ("outside therapy") performed with the paralyzed arm during the planned study - including baseline and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-07; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer Assessment Scale | four and one weeks prior to intervention, four weeks after intervention started, at the end of intervention(eight weeks), two months and six months follow-up

SECONDARY OUTCOMES:
Wolf Motor Function Test, Stroke Impact Scale, Motor Activity Log, modified Ashworth Scale, abnormal joint synergies, active range of motion (ROM), muscle strength, and spatial precision of hand positioning. | three and one weeks prior to intervention, four weeks after intervention started, at the end of intervention(eight weeks), two months and six months follow-up
fMRI | before and after 8 weeks therapy, 2-months follow-up
  in 20 Patients fMRI will be recorded while patients interact with an MR-compatible manipulandum

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof., Study Director — Sensory Motor Systems Lab, ETH Zürich; Armin Curt, Prof., Principal Investigator — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Nef T, Mihelj M, Riener R. ARMin: a robot for patient-cooperative arm therapy. Med Biol Eng Comput. 2007 Sep;45(9):887-900. doi: 10.1007/s11517-007-0226-6. Epub 2007 Aug 3. PMID 17674069
- [Derived] Valero-Cuevas FJ, Klamroth-Marganska V, Winstein CJ, Riener R. Robot-assisted and conventional therapies produce distinct rehabilitative trends in stroke survivors. J Neuroeng Rehabil. 2016 Oct 11;13(1):92. doi: 10.1186/s12984-016-0199-5. PMID 27724916
- [Derived] Klamroth-Marganska V, Blanco J, Campen K, Curt A, Dietz V, Ettlin T, Felder M, Fellinghauer B, Guidali M, Kollmar A, Luft A, Nef T, Schuster-Amft C, Stahel W, Riener R. Three-dimensional, task-specific robot therapy of the arm after stroke: a multicentre, parallel-group randomised trial. Lancet Neurol. 2014 Feb;13(2):159-66. doi: 10.1016/S1474-4422(13)70305-3. Epub 2013 Dec 30. PMID 24382580